CLINICAL TRIAL: NCT04319549
Title: Post Operative Pain and Expression of Substance P, IL8 After the Use of Ketorolac Irrigant Following Single Visit Root Canal Treatment
Brief Title: Ketorolac Irrigant on Post Operative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nasrin Salem Bazina, principal invistigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ketorolac irrigant
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-03

CONDITIONS: Acute Irreversible Pulpitis With Apical Periodontitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 ketorolac tromethamine irrigant (Experimental): group 1 patients with acute irreversible pulpitis with apical periodontitis
  Interventions: Other: Ketorolac Tromethamine irrigant
- group 2 sodium hypochlorite irrigant (Active Comparator): group 2 patients with acute irreversible pulpitis with apical periodontitis
  Interventions: Other: sodium hypochlorite irrigant

INTERVENTIONS:
Other: Ketorolac Tromethamine irrigant — Ketorolac tromethamine, a potent NSAID available in both oral and injectable forms, is over 400 times more potent as a selective inhibitor of COX-1 over COX-2 than many other drugs. When ketorolac tromethamine was used as an intracanal medicament in teeth with irreversible pulpitis undergoing root canal treatment, it contributed to significant post operative pain relief.
  Arms: group 1 ketorolac tromethamine irrigant
Other: sodium hypochlorite irrigant — NaOCl is the gold standard and the most commonly used root canal irrigant. NaOCl is able to dissolve the organic tissues inside root canal due to its alkalinity (pH11), which causes amino acid degradation and hydrolysis through the production of chloramine molecules. In addition, it possesses highly antibacterial effect and its low cost makes it the most frequently used root canal irrigant. Dual rinse is considered an effective time saving root canal irrigant with a better antibacterial property in comparison to NaOCl alone. In addition to its effectiveness on smear layer removal and reduction in the debris accumulation during root canal instrumentation.
  Arms: group 2 sodium hypochlorite irrigant

SUMMARY:
Endodontic post-treatment pain management is one of the most challenging problems in the clinical practice of endodontics. Although this pain is decreased after root canal treatment, there may be residual symptoms due to inflammation. It has been reported that up to 80% of patients with preoperative pain, will report pain after endodontic treatment, which might range from mild to severe. Management of endodontic pain should involve all steps of treatment including preoperative pain control through accurate diagnosis and reduction of anxiety, intraoperative pain control through effective and profound local anesthetic, operative techniques and that can be achieved through a variety of pharmacologic agents. Many mechanisms have been proposed to explain the reason for postoperative pain including the sensitization of nociceptors by inflammatory mediators. Among these chemical inflammatory mediators are the prostaglandins which is the terminal product of arachidonic acid metabolism, through the cyclooxygenase (COX) pathway. Endodontic treatment can cause the release of inflammatory mediators (e.g. prostaglandins, leukotrienes, bradykinin, platelet- activating factor and substance P) into the surrounding periapical tissues, causing pain fibers to be directly stimulated (by bradykinin for instance) or sensitized (by prostaglandins). In addition, the vascular dilation and increased permeability as a consequence of periradicular inflammation, cause edema and increased interstitial tissue response. Single-visit root canal treatment is common in some endodontic practices. However, one of the main concerns with this approach has been the fear of post- operative pain. Mechanical, chemical and microbiological injuries to the peri- radicular tissues during root canal treatment have been suggested as possible causes of post-operative pain. The role of irrigating solutions used during root canal treatment to help control post-operative pain is unclear. While certain studies have observed a reduction in post-operative pain with particular types and concentrations of irrigating solutions, other studies have reported no difference in post-operative pain with the different irrigating solutions .

DETAILED DESCRIPTION:
When the treatment itself appears to initiate the onset of pain and/or swelling, the result can be very distressing to both the patient and the operator.

Patients might even consider postoperative pain and flare-up as a benchmark against which the clinician's skills are measured. Prevalence of postoperative pain or flare-up is, therefore, one of the influencing factors when making a clinical decision. Better management of postoperative pain increases the patients' confidence in dentist's skills and gives positive attitude toward dental profession. The major cause of this pain is thought to be because of the release of inflammatory mediators that stimulate sensitive nociceptors surrounding the tooth. The resultant stimulation of both central and peripheral mechanisms is described as hyperalgesia which is defined as an increase in the perceived degree of a painful stimulus. One of the many inflammatory mediators, IL-8 has been extensively considered as a potential marker for irreversible pulpitis. Increased expression of IL-8 is correlated with increased polymorphonuclear neutrophils (PMNs) within the pulp because IL-8 induces neutrophil chemotaxis and release of degradation enzymes during degranulation. Substance P was the initial neuropeptide identified in the dental tissues. The released substance P further promotes the release of short-lived inflammatory mediators providing a fresh supply of prostaglandins (iPGE2), leukotriene (iLTB4) and bradykinins. These sustained effects of the released inflammatory mediators are part of a local positive feedback cycle. Neuronal responses in the dental pulp due to caries have been shown to alter the anatomical distribution of nerve fibers, leading to increases in neuropeptide expression and increased pain sensitivity as a result of peripheral sensitization. Prostaglandin construction in this inflammatory process is via the cyclooxygenase pathway. Ketorolac tromethamine, a potent NSAID available in both oral and injectable forms, is over 400 times more potent as a selective inhibitor of COX-1 over COX-2 than many other drugs. When ketorolac tromethamine was used as an intracanal medicament in teeth with irreversible pulpitis undergoing root canal treatment, it contributed to significant post operative pain relief.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 15-60 years old.
2. Systemically healthy patient (ASA I or II).
3. Male & female.
4. Molar or premolar teeth with:
5. Preoperative moderate to severe pain.
6. with or without slight widening in the periodontal membrane space
7. Patients' acceptance to participate in the trial.

Exclusion Criteria:

1. Patients allergic to anesthetics.
2. Patients having significant systemic disorder (ASA III or IV).
3. Hemostatic disorders or anti-coagulant therapy during the last month.
4. Retreatment cases
5. Pregnant women: Avoid radiation exposure, anesthesia, and medication.
6. No restorability: Hopeless tooth.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
post operative pain | intensity of pain by categorical scale from 1-4
  post operative pain will be measured by categorical scale

SECONDARY OUTCOMES:
substance P,IL8 Level | baseline
  inflammatory mediator will be measured by ELISA

REFERENCES:
- [Background] Bamini L, Anand Sherwood I, Abbott PV, Uthandakalaipandian R, Velu V. Influence of anti-inflammatory irrigant on substance P expression for single-visit root canal treatment of teeth with irreversible pulpitis. Aust Endod J. 2020 Apr;46(1):73-81. doi: 10.1111/aej.12353. Epub 2019 Jul 3. PMID 31270901
- [Background] Evangelin J, Sherwood IA, Abbott PV, Uthandakalaipandian R, Velu V. Influence of different irrigants on substance P and IL-8 expression for single visit root canal treatment in acute irreversible pulpitis. Aust Endod J. 2020 Apr;46(1):17-25. doi: 10.1111/aej.12340. Epub 2019 Jul 3. PMID 31270902